CLINICAL TRIAL: NCT04815642
Title: Retrospective Study Evaluating Hypofractionated Radiotherapy Concomitantly With Weekly Boost for Breast Cancer Patients Treated With Conservative Breast Surgery
Brief Title: Hypofractionated Radiotherapy Concomitantly With Weekly Boost for Breast Cancer Patients Treated With Conservative Breast Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada mohamed shawky, Principal investigator, Assiut University
Other Study IDs: Radiation in breast cancer
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiotherapy — Hypofractionated radiotherapy concomitantly with weekly boost

SUMMARY:
This is a retrospective study on evaluation of the efficacy and the safety of a hypofractionated radiotherapy course with weekly concomitant boost for breast cancer patients treated with conservative breast surgery .

ELIGIBILITY:
Inclusion Criteria:

1. women aged from 18 and up to 55 years old.
2. Histologically diagnosed with breast carcinoma (ductal and others )
3. All patients with conservative breast surgery.
4. Including all patients with in all stages except those stage IV.
5. All patients with clear free surgical margin.
6. patients received hypofractionated radiotherapy with weekly concomitant boost

Exclusion Criteria:

1. Evidence of distant metastatic deposites.
2. patients with mastectomy
3. patients with prior irradiation to thoracic region.
4. pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Efficacy of a short accelerated hypofractionated radiotherapy course with once weekly concomitant photon boost for women patients diagnosed with breast cancer and treated with conservative breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | baseline
  Disease Free survival

REFERENCES:
- [Background] 1. Ferlay J, Soerjomataram I, Dikshit R, et al. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J cancer. 2015;136(5):E359-386. 2. L. A. Torre, F. Bray, R. L. Siegel, J. Ferlay, J. Lortet-Tieulent, and A. Jemal, "Global cancer statistics, 2012," CA. Cancer J. Clin., vol. 65, no. 2, pp. 87-108, Mar. 2015. 3. A. S. Ibrahim, H. M. Khaled, N. N. Mikhail, H. Baraka, and H. Kamel, "Cancer incidence in egypt: results of the national population-based cancer registry program.," J. Cancer Epidemiol.,vol. 2014, p. 437971, Sep. 2014. 4 Tamer M Samy , Samia Abdelkareem , Marwa Abdelgawad , Shimaa Ahmed ..Cardiac toxicity of hypofractionated radiotherapy in left breast cancer 1221 1 Radiation Oncology, South Egypt Cancer Institute (SECI), Asyut University, Egypt. 2 Clinical Oncology, Faculty of Medicine, Asyut University, Egypt.2018 5.Darby S. McGale P.Correa C.et al. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10, 801 women in 17 randomised trials. Lancet. 2011; 378: 1707-1716 View in Article 6.van Werkhoven E.Hart G.van Tinteren H.et al. Nomogram to predict ipsilateral breast relapse based on pathology review from the EORTC 22881-10882 boost versus no boost trial. Radiother Oncol. 2011; 100: 101-107 7.-Bartelink H.Maingon P.Poortmans P.et al. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015; 16: 47-56 8 Darby S, McGale P, Correa C, Taylor C, Arriagada R, et al..Early Breast Cancer Trialists' Collaborative G, Effect of radiotherapy after breast- conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011;378(9804):1707-16. 10.1016/S0140-6736(11)61629-2 9.Hughes KS, Schnaper LA, Bellon JR, Cirrincione CT, Berry DA, McCormick B, et al. Lumpectomy plus tamoxifen with or without irradiation in women age 70 years or older with early breast cancer: long-term follow-up of CALGB 9343. Journal of clinical oncology: official journal of the American Society of Clinical Oncology. 2013;31(19):2382-7. 10.Interdisziplinäre S3-Leitlinie für die Früherkennung, Diagnostik, Therapie und Nachsorge des Mammakarzinoms [Internet]. 2017. 11.Bartelink H, Maingon P, Poortmans P, et al. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol 2015; 16: 47-56. 12.Vrieling C, van Werkhoven E, Maingon P, et al. Prognostic factors for local control in breast cancer after long-term follow-up in the EORTC boost vs no boost trial: a randomized clinical trial. JAMA Oncol 2017; 3: 42-48. 13.Jones HA, Antonini N, Hart AA, et al. Impact of pathological characteristics on local relapse after breast-conserving therapy. J Clin Oncol. 2009;27(30):4939-4947.PubMedGoogle ScholarCrossref 14.Bartelink H, Maingon P, Poortmans P, et al; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer. Lancet Oncol. 2015;16(1):47-56. 15.Cox JD et al. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC ); Int J Radiat Oncol Biol Phys.1 995 Mar 30 ;31 (5):1341-6.